CLINICAL TRIAL: NCT02187510
Title: Umbilical Cord Milking Compared With Delayed Cord Clamping to Increase Plancental Transfusion in Preterm Infants Less Than 34 Weeks' Gestation Born by Cesarean Section. Randomised Clinical Trial
Brief Title: Umbilical Cord Milking vs Delayed Cord Clamping in Preterm Infants Born by Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Mònica Domingo Puiggròs, Medical Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSPTNeonat2014_01
Record Dates: First submitted 2014-06-06; First posted 2014-07-11 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Premature Infant; Umbilical Cord; Milking; Delayed Clamping
Keywords: Hemodynamics; Premature Infant; Umbilical cord; Milking; Delayed clamping
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umbilical cord milking (Experimental): Once the preterm is born keep the baby from the mother's thighs. The obstetrician cord milking three times (2seconds/milking) taking the cord from the base 20cm respect towards the baby. Then clamp de cord.
  Interventions: Procedure: Umbilical cord milking
- Delayed cord clamping (Active Comparator): Once the preterm is born the neonatologist keep the baby beside the mother at level of the operating table during 30 seconds without cord clamping. The baby is covered with a polythene bag and put a cap on his head. Then the obstetritian clamp the cord.
  Interventions: Procedure: Delayed cord clamping

INTERVENTIONS:
Procedure: Umbilical cord milking — Once the preterm is born keep the baby from the mother's thighs. The obstetrician cord milking three times (2seconds/milking) taking the cord from the base 20cm respect towards the baby. Then clamp de cord.
  Arms: Umbilical cord milking
Procedure: Delayed cord clamping — Once the preterm is born the neonatologist keep the baby beside the mother at level of the operating table during 30 seconds without cord clamping. The baby is covered with a polythene bag and put a cap on his head. Then the obstetritian clamp the cord.
  Arms: Delayed cord clamping

SUMMARY:
The purpose of this study is to determine whether the umbilical cord milking in preterm infants born by cesarian section less than 34 weeks is more effective than delayed cord clamping to obtain higher levels of hemoglobin.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 34 weeks' gestation born by cesarean section

Exclusion Criteria:

* Inability to obtain informed consent from the mother state
* Monochorionic-monoamniotic twin gestation
* Placenta abruption
* Uterine rupture
* Transplacental cesarean
* Hydrops fetalis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Haemoglobin | 1 hour and 24 hours at born
  g/dl

SECONDARY OUTCOMES:
Apgar Score | 1 and 5 minutes
  Basic score to mesure the newborn status. From 0 to 10.
Arterial pressure | 2, 6, 12, 24, 36 and 48 hours of life
  Mean of systolic and dyastolic arterial pressure in mm Hg
Orine volume | 24 and 48 hours of life
  Total volume of orine at 24 and 48 hours of life. Total ml.
Use of vasopresors drugs | 24 hours of life
  To use or not to use the vasopresors drugs during the first 24 hours of life
Number of concentrate hematies transfusion | participants will be followed for the duration of hospital stay (from 2 weeks up to 3 months)
  Total number of concentrate hematies transfusions during the hospital stay. The stay should vary depending of the gestacional age, from 2 weeks up to 3 months.
Intraventricular hemorrhage | participants will be followed for the duration of hospital stay (from 2 weeks up to 3 months)
  Presence of intraventricular hemorrhage mesured by cerebral ultrasound Degree of the hemorrhage by Papile
Bronchopulmonary dysplasia | participants will be followed for the duration of hospital stay (from 2 weeks up to 3 months)
  Presence of Bronchopulmonary dysplasia and the degree, mesured by Spanish classification (M. Sanchez Luna)
Total intensive care unit stay | Participants will be followed for the duration of hospital stay (from 2 weeks up to 3 months)
  Mesured in days. The stay should vary depending of the gestacional age, from 2 weeks up to 3 months.
Hematocrit | 1 hour and 24 hours at born
  In percentage

CONTACTS AND LOCATIONS:
Overall Officials: Monica Domingo-Puiggros, MD, Study Director — Corporacio Sanitaria Parc Tauli
Locations (1):
- Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona, Spain